CLINICAL TRIAL: NCT02384161
Title: Exercise Intermittent Isometric Handgrip Associated With Different Levels of External Vascular Compression: Acute Effects on Neuromuscular Response
Brief Title: Exercise Intermittent Isometric Handgrip and Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Mikhail Santos Cerqueira, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UFPernambucoMK
Record Dates: First submitted 2015-02-23; First posted 2015-03-10 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Total RBF + Exercise Isometric (Experimental): Volunteers will undergo a year of intermittent isometric handgrip (intervention) in the dominant member associated with a total obstruction of blood flow, which will be conducted through a "cuff" pressure applied to the proximal region of the dominant limb.
  Interventions: Other: Isometric exercise Intermittent
- Partial RBF + Exercise Isometric (Experimental): Volunteers will undergo a year of intermittent isometric handgrip (intervention) in the dominant member associated with a partial obstruction of blood flow, which will be conducted through a "cuff" pressure applied to the proximal region of the dominant limb.
  Interventions: Other: Isometric exercise Intermittent
- Free BR + Exercise Isometric (Placebo Comparator): Volunteers will undergo a year of intermittent isometric handgrip (intervention) in the dominant limb with the free blood flow. A 'cuff' pressure on the member of the proximal region, but with a pressure that will not interfere with blood flow will be applied.
  Interventions: Other: Isometric exercise Intermittent

INTERVENTIONS:
Other: Isometric exercise Intermittent — Intermittent isometric exercise is characterized by an interval muscle contraction (one period and another relaxed contracted period) in which there is no generation of voltage change in the length of the muscle fiber.

SUMMARY:
Isometric handgrip exercises are used to explain the effects of fatigue on the strength and activation of the muscles involved. Blood flow available at the time of exercise can influence this fatigue process, as some studies demonstrate changes in the pattern of muscle recruitment and strength recovery when the exercise is performed in combination with an external total obstruction (through a pressure cuff or tourniquet ) blood flow. Low intensity exercises associated with external partial obstruction of blood flow has been widely used and studied, mainly due to its effect on increasing strength and muscle hypertrophy, often comparable to those observed in conventional exercises (ie, without external obstruction of blood flow) High intensity. Despite the vast literature on this method, some topics need to be better informed about the underlying neuromuscular physiology to such effects (strength and hypertrophy) and the process of fatigue during isometric exercises associated with partial obstruction of blood flow. The aim of this study is to evaluate the acute effects on neuromuscular response in healthy adults undergoing an intermittent isometric exercise protocol with different levels of external compression. In a study of the "crossover" male volunteers will be submitted to three intermittent isometric exercise protocols (with a load of 45% of maximum voluntary isometric strength) associated with three different levels of obstruction (held by a pressure cuff) blood flow (total obstruction, partial obstruction and free blood flow). The protocols will be performed on three different days (with a minimum of 48 hours between them). Will be considered as acute neuromuscular responses spending time to failure in the task, the electromyographic activity of the flexor muscles of the wrist and fingers, and the recovery curve of maximum voluntary isometric strength after exercise. The main hypothesis of this study is that exercise is performed when associated with partial obstruction of blood flow, the time spent until the failed job is similar to that seen when exercise is performed with free blood flow, and the recovery of strength and electromyographic activity will be similar to that observed in the exercise associated with total obstruction of blood flow.

DETAILED DESCRIPTION:
Muscle fatigue is a process widely disbelieved and studied in the literature. Isometric handgrip exercises have been widely utilized to explain the effects of fatigue on the strength and activation of the muscles involved in certain exercises. Among the many factors that can influence the process of muscular fatigue, blood flow available at the time of exercise is an aspect of fundamental importance, as some studies demonstrate changes in the pattern of muscle recruitment and strength recovery when the exercise is performed associated with an external obstruction of blood flow.

Resistance exercise associated with partial obstruction of blood flow (ischemic exercise) is gaining notoriety in the scientific environment, mainly due to strong evidence indicating that such activity can increase strength and muscle hypertrophy, even when performed with low intensity loads. The underlying neuromuscular mechanisms such effects are still partially unknown, and some studies have shown differences in the recruitment of motor units during its execution, and the relationship fatigue-strength after ischemic resistance exercise. Nevertheless, there are still some gaps in the literature regarding the neuromuscular responses during and after unilateral intermittent isometric handgrip protocols to failure in the associated task to partial obstruction of blood flow.

Evidence suggests that the total obstruction of blood flow decreases performance and accelerates the recovery of the isometric strength after fatigue protocols, but the effects of partial obstruction on these variables remain unknown. In the above so far, it seems that isometric fatigue protocols associated with remote obstruction (away from the venue of the exercise) blood flow can influence acutely in strength members at a distance, but it is not known as a protocol unilateral isometric fatigue associated with partial and complete obstruction of blood flow can influence acutely the strength of the contralateral limb (ie, not subject to any type of exercise). Thus, the realization of this study is justified by the possibility of answering these questions still little studied, with regard to neuromuscular factors of ischemic resistance training.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers classified as irregularly active or active
* Volunteers ranked within the normal range (18.5 to 24.9 kg / m2), the Body Mass Index (BMI).

Exclusion Criteria:

* Smokers volunteers will be excluded, that are using vasoactive drugs and having fracture history in upper limbs; hypertension, venous insufficiency, cardiac insufficiency or any other cardiovascular disease; epilepsy, stroke or some other neurological disease or any other condition that prevents you from performing the exercise protocol.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary isometric strength. | 3 months
  Recovery of maximal voluntary isometric strength in the dominant member.
Time to task failure. | 3 months
  Recovery of time to task failure in the dominant member.
electromyography activity. | 3 months
  Recovery electromyographic activity in the dominant member.

SECONDARY OUTCOMES:
Contralateral maximum voluntary isometric strength (non-dominant limb). | 3 months
  Contralateral maximum voluntary isometric strength (non-dominant limb).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil